CLINICAL TRIAL: NCT07406568
Title: Move Healthier Group
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth.W.Lampe, Clinical Psychology Fellow, Weight Center, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02003218
Record Dates: First submitted 2026-01-13; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Overweight
Keywords: exercise; physical activity; disordered eating; eating disorder
MeSH Terms: conditions — Obesity; Overweight; Motor Activity; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Move Healthier Group Intervention Arm (Experimental): This group-based intervention aims to promote healthy exercise without increasing risk for compensatory exercise or other disordered eating behaviors. Participants will attend 12 weekly 90-minute group intervention sessions via telehealth software.
  Interventions: Behavioral: Move Healthier Intervention

INTERVENTIONS:
Behavioral: Move Healthier Intervention — The intervention aims to increase exercise using cognitive and behavioral skills integrated across several treatment manuals including the Physical Activity Cognitively Enhanced (PACE) intervention for healthy exercise promotion in eating disorders, acceptance-based and standard behavioral weight loss manuals, and affect-guided exercise prescriptions.

SUMMARY:
The researchers are developing a new exercise-focused group and are interested in studying whether this group helps people increase their exercise without increasing risk for disordered eating behaviors.

DETAILED DESCRIPTION:
Individuals seeking weight loss are often encouraged to increase their exercise engagement as a health-promoting behavior. However, exercise engagement is often connected directly to caloric intake within weight loss interventions, so it is likely that individuals seeking weight loss are engaging in some level of compensatory exercise even in the absence of other disordered eating symptoms. Compensatory exercise is defined as exercising to "offset" or "make up for" calories consumed with the intent of controlling one's body weight or shape. The researchers are developing a new group to promote healthy exercise and are interested in studying whether this group helps people increase their exercise without increasing risk for compensatory exercise or other disordered eating behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Seen for weight loss treatment at DHMC Weight Center within the past year
* Speak, read, & write English fluently
* Age 18 or older
* Appropriate for group visits (as assessed by referring provider)

Exclusion Criteria:

* Meets DSM-5 criteria for an eating disorder based on behavior frequencies reported on baseline EDE-Q
* Report contraindications for unsupervised physical activity on the PAR-Q, or have not been medically cleared by an MD for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Objective physical activity | From enrollment to the end of treatment at 12 weeks
  Objective physical activity will be measures as the total number of minutes per week of physical activity measured via Fitbit device worn during waking hours. The Fitbit data will yield a total count of the number of minutes of moderate-to-vigorous physical activity for each week during the intervention period, with higher counts indicating greater levels of activity.
Self-reported physical activity | From enrollment to the end of treatment at 12 weeks
  Participants will also complete self-report measures of physical activity, including the International Physical Activity Questionnaire (IPAQ) and IPAQ-short form at group sessions and study assessments. The IPAQ asks patients to report on their total physical activity engagement over the past 7 days by light, moderate, and vigorous activity categories. The IPAQ yields a total count of the number of minutes of moderate-to-vigorous physical activity over the past week, with higher minutes indicating more activity.
Eating disorder symptoms | Baseline and post-intervention (week 12)
  ED symptoms will be assessed via the Eating Disorder Examination Questionnaire (EDE-Q 6.0), which asks about ED symptoms over the past month (28 days). Compensatory exercise engagement will be assessed via an item asking, "Over the past 28 days, how many times have you exercised to "make up for" a binge-eating episode, and compulsive exercise will be assessed using the item "...how many times have you felt driven/compelled to exercise?" EDE-Q items are averages to calculate a total score ranging from 0-6, with higher scores indicating higher levels of eating pathology.

SECONDARY OUTCOMES:
Weight bias internalization | baseline and post-intervention (week 12)
  Internalized weight stigma will be measured using the Weight Bias Internalization Scale (WBIS). The WBIS comprises 11 items measuring self-directed weight bias and has shown excellent convergent and divergent validity within the population of interest. The WBIS items are averaged to yield a total score ranging from 1-7, with higher scores reflecting higher internalized weight bias.
intervention acceptability | post-intervention (week 12)
  Participants will complete qualitative interviews at post-treatment to provide feedback on group format, acceptability, utility, etc. Qualitative analysis of these interview transcripts will elucidate themes related to group acceptability.
intervention feasibility | post-intervention (week 12)
  Feasibility will be measured via group attendance rates across the 12 sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Salwen-Deremer, PhD, Study Director — Dartmouth Health; Elizabeth Lampe, PhD, Principal Investigator — Dartmouth Health
Locations (1):
- Dartmouth-Hitchcock Clinics, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared to facilitate future research study recruitment and/or to answer future research questions. There is no plan to share IPD at this time.